CLINICAL TRIAL: NCT00883064
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Eon Labs Manufacturing Inc. (USA) and Zeneca (USA) (Zestril) 40 mg Lisinopril Tablet Administered as a 1 x 40 mg Tablet in Health Adult Males Under Fasting Conditions.
Brief Title: To Demonstrate the Relative Bioequivalence of Lisinopril 1 x 40 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00102
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Lisinopril; Tablets

ARMS (2):
- 1 (Experimental): Lisinopril 40 mg Tablet (EON Labs Manufacturing Inc, USA)
  Interventions: Drug: Lisinopril 40 mg Tablet (EON Labs Manufacturing Inc, USA)
- 2 (Active Comparator): Lisinopril 40 mg Tablet (Zestril) (Zeneca, USA)
  Interventions: Drug: Lisinopril 40 mg Tablet (Zestril) (Zeneca, USA)

INTERVENTIONS:
Drug: Lisinopril 40 mg Tablet (EON Labs Manufacturing Inc, USA)
  Arms: 1
Drug: Lisinopril 40 mg Tablet (Zestril) (Zeneca, USA)
  Arms: 2

SUMMARY:
To Demonstrate the Relative Bioequivalence of Lisinopril 1 x 40 mg Tablets Under Fasting Conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2000-03; Primary Completion 2000-04 (Actual); Study Completion 2000-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 23 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Masson, Pharm.D., Principal Investigator — Anapharm